CLINICAL TRIAL: NCT04478097
Title: A Randomized, Open, Single-dose, 3 Period Partial Replicated Crossover-design Clinical Trial to Evaluate the Safety and Pharmacokinetic Characteristics After Administration of CKD-333 or Co-administration of CKD-330 and D086 in Healthy Volunteers Under Fasting Conditions
Brief Title: Clinical Trial to Evaluate the Safety and Pharmacokinetic Characteristics in Healthy Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A70_09BE2005
Record Dates: First submitted 2020-07-17; First posted 2020-07-20 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Reference-Reference-Test (Experimental)
  Interventions: Drug: CKD-330 Tab. and D086 Tab.; Drug: CKD-333 Tab.
- Reference-Test-Reference (Experimental)
  Interventions: Drug: CKD-330 Tab. and D086 Tab.; Drug: CKD-333 Tab.
- Test-Reference-Reference (Experimental)
  Interventions: Drug: CKD-330 Tab. and D086 Tab.; Drug: CKD-333 Tab.

INTERVENTIONS:
Drug: CKD-330 Tab. and D086 Tab. — 1T
  Other Names: Reference
Drug: CKD-333 Tab. — 1T
  Other Names: Test

SUMMARY:
This study is a randomized, open, single-dose, 3 period partial replicated crossover-design study to investigate the pharmacokinetic profiles and safety of CKD-333 in healthy volunteers.

DETAILED DESCRIPTION:
To healthy subjects of fifty-one (51), following treatments are administered dosing in each period and wash-out period is a minimum of 14 days.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults over the age of 19 years and under the age of 55 years at the time of screening
2. Individuals who had 17.5 kg/m2 ≤ Body Mass Index(BMI) < 30.5kg/m2 and men's total body weight ≥ 55 kg, women's total body weight ≥ 45 kg

   * BMI = Weight(kg)/ Height(m)2
3. Individuals without congenital/chronic diseases and without abnormal symptoms or diagnosis based on a medical examination within the last 3 years
4. Individuals who were deemed to be appropriate as study subjects following laboratory tests (hematology, blood chemistry, urinalysis, viral/bacterial, etc.) and vital signs, ECG etc. performed at screening
5. Individuals who signed an informed consent form and decided to participate in the study after being fully informed of the study prior to participation
6. Individuals who agreed proper contraception during the study and did consent to not donation of sperm 1 month after the last dose of study drug infusion
7. Individuals with the ability and willingness to participate the entire study period

Exclusion Criteria:

1. Individuals with a medical evidence or a history of clinically significant hepatobiliary, renal, neurologic, respiratory, digestive, endocrine, blood-oncology, urinary, cardiovascular, musculoskeletal or psychiatric
2. Individuals with a medical history of gastrointestinal disease (e.g., Crohn's disease and ulcer) or gastrectomy (excluding simple appendectomy or herniotomy) that may affect drug absorption
3. Individuals with the following results at screening test:

   * ALT or AST > 2x the upper limit of the normal range
   * Creatinine > upper limit of the normal range or eGFR with MDRD <60 ml/min/1.73 m2
   * ECG Result, QTc > 450msec
   * CPK > UNL(upper normal limit) x 3.0
   * K > 5.5mEq/l
   * Hct < lower limit of the normal range
4. A history of regular alcohol consumption exceeding 21 units/week within the 3 months(1 unit = 10 g = 12.5 ml) prior to screening or individuals who cannot quit drinking from 48hr prior to the first dose to end of last blooding (1 drink (250 mL) of beer (5%) = 10 g; 1 drink (50 mL) of hard liquor (20%) = 8 g; 1 drink (125 mL) of wine (12%) = 12 g)
5. Individuals who smoked more than 20 cigarettes per day within 6 months prior to screening or cannot quit smoking during hospitalization period
6. Individuals who had been administered investigational product(s) of other clinical study or bioequivalence study within the 6 months prior to the first dose of this study
7. Following vital signs results at screening

   * Sitting systolic blood pressure ≥ 140 mmHg or < 90 mmHg
   * sitting diastolic blood pressure ≥90 mmHg or <60 mmHg
8. Individuals with a medical history of significant drug abuse within one year prior to the screening or positive for abuse drug in urine test results at screening
9. Individuals taking medication known to significantly induce or inhibit drug metabolizing enzymes within 30days before the first administration of clinical trial drug
10. Individuals who had taken prescription or nonprescription drugs within the 10 days prior to the first dose of investigational product(s)
11. Individuals who donated whole blood within the 2 months, or blood components within 1 month prior to the first dose of the investigational product(s)
12. Individuals with hypersensitivity to investigational products or the investigational products ingredients
13. Patients or conditions deemed to be at risk for using investigational products

    * Patient with hyperkalemia
    * Patients with hepatopathy
    * Patients with hereditary angioedema, ACE inhibitors or angiotensin 2 receptor antagonists who have a history of angioedema
    * Primary hyperaldosteronism
    * Patients with aortic valve stenosis, mitral (valve) stenosis, hypertrophic obstructive cardiomyopathy
    * Patients with ischemic heart disease, ischemic cardiovascular disease, cerebrovascular disease
    * Patients with Intravascular volume depletion
    * Patients with diabetes or kidney failure
    * Patients with renal artery stenosis
    * Patients with muscle disease
    * Patients with Hypothyroidism
    * Patients with a history of muscle toxicity when using statins or fibrates
    * Patients who have recently had a kidney transplant
    * Patients with history of shock
14. Individuals with hereditary diseases of galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption etc.
15. Individuals who drunk grapefruit juice or caffeine more than 5 cup per day within 3 months prior to screening or cannot quit drinking during clinical trials period
16. Individuals who cannot eat standard meal in institution
17. Women who are pregnant or may be pregnant
18. Individuals who were deemed to be inappropriate to participate in the study by the investigator

Ages: 19 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Estimated)
Dates: Start 2020-07-14 (Estimated); Primary Completion 2020-11-05 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
AUCt of CKD-330, D086, CKD-333 | [Time Frame: Pre-dose (0 hour), post-dose 0.17, 0.33, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48, 72 hours]
  Area under the CKD-330/D086/CKD-333 concentration in blood-time curve from zero to final
Cmax of CKD-330, D086, CKD-333 | [Time Frame: Pre-dose (0 hour), post-dose 0.17, 0.33, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48, 72 hours]
  The maximum CKD-330/D086/CKD-333 concentration in blood sampling time t

CONTACTS AND LOCATIONS:
Locations (1):
- Jang Hee Hong, Daejeon, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim JH, Song JH, Kim M, Hong JH, Sunwoo J, Jung JG. Pharmacokinetic Comparison of a Fixed-Dose Combination of Candesartan Cilexetil/Amlodipine/Atorvastatin Versus Co-administration of Individual Formulations in Healthy Participants. Adv Ther. 2024 Jul;41(7):2808-2825. doi: 10.1007/s12325-024-02869-y. Epub 2024 May 21. PMID 38771476